CLINICAL TRIAL: NCT03909581
Title: Randomized Study Of Endoscopic Coronary Arterial Bypass Versus Percutaneous Coronary Intervention for Left Anterior Descending Artery Revascularization
Brief Title: EndoACAB vs PCI for LAD Revascularization
Acronym: ENPILА
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center of Surgery, Russia (Other Government)
Responsible Party: Principal Investigator, Vadim Popov, M.D., Ph.D, Prof. Head of cardiovascular Department, National Research Center of Surgery, Russia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7t7sci9q
Record Dates: First submitted 2019-02-26; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases; Myocardial Ischemia
Keywords: CABG; EndoCAB; PCI
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic coronary arterial bypass (Active Comparator): is defined, for the purposes of this trial, as a planned off-pump minimally invasive (sternal-sparing), isolated LIMA-LAD revascularization
  Interventions: Procedure: Endoscopic coronary arterial bypass
- Percutaneous Coronary Intervention (Active Comparator): will be performed using standard techniques at the discretion of the operator
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Endoscopic coronary arterial bypass — is defined, for the purposes of this trial, as a planned off-pump minimally invasive (sternal-sparing), isolated LIMA-LAD revascularization (50 participants)
  Other Names: EndoCAB
  Arms: Endoscopic coronary arterial bypass
Procedure: Percutaneous Coronary Intervention — will be performed using standard techniques at the discretion of the operator (50 participants)
  Other Names: PCI
  Arms: Percutaneous Coronary Intervention

SUMMARY:
The purpose of this study is to determine which treatment option is better for patients who have isolated coronary artery disease (blockages of one vessel supplying blood to the heart muscle). The treatment options compared in this study are:

1. Endoscopic coronary arterial bypass
2. Percutaneous Coronary Intervention. This study is aimed to determine the best treatment for patients with coronary artery disease.

DETAILED DESCRIPTION:
Coronary artery disease (CAD), also known as coronary heart disease (CHD) involves the progressive narrowing of the arteries that nourish the heart muscle. CAD is the main cause of death in Russia.

Patients with LAD disease have worse coronary flow outcomes Currently established types of myocardial revascularization are coronary artery bypass grafting (CABG) and percutaneous coronary interventions (PCI). High effectiveness of CABG was proved by multiple studies. PCI is a first line therapy in the treatment of one vessel disease due to the less invasive approach and current technological possibilities of this revascularization method.

However, the established gold standard of multivessel coronary blockage treatment is CABG. It was reflected in the latest ESC/EACTS Guidelines on Myocardial Revascularization, due to the better early and late outcomes associated with the graft specifics.

On the other hand, standard CABD operation has a high injury and morbidity rate, which were factors for development of less invasive techniques of CABG.

According to the latest ESC/EACTS guidelines there are no advantages between PCI and CABG in the LAD disease treatment, both methods are Class I; level of evidence A.

The choice between myocardial revascularization methods in patients with LAD disease is the critical task.

ELIGIBILITY:
Inclusion Criteria:

* The presence of isolated lesions of LAD are available for revascularization PCI and EndoCAB
* Suitable candidate for both PCI and EndoCAB as determined by clinical assessment and angiogram review by an interventional cardiologist and a cardiac surgeon at the enrolling clinical site
* Age ≥ 18 years

Exclusion Criteria:

* Previous cardiac surgery of any kind, including CABG
* Previous thoracic surgery involving the left pleural space
* Need for concomitant vascular or other cardiac surgery during the index hospitalization (including, but not limited to, valve surgery, aortic resection, left ventricular aneurysmectomy, and carotid endarterectomy or stenting)
* Indication for chronic oral anticoagulation therapy at the time of randomization
* Extra-cardiac illness that is expected to limit survival to less than 5 years
* Allergy or hypersensitivity to any of the study drugs or devices used in the trial
* Therapy with an investigational drug, device or biologic within 1 year prior to randomization, or plan to enroll patient in additional investigational study during participation in this trial
* Unable to give informed consent or potential for noncompliance with the study protocol in the judgment of the investigator
* Ejection fraction of 40% or less Left ventricular dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
MACCE | 1 year
  Major adverse cardiac and cerebral events (MACCE), including death,a composite of major cardiac and cerebrovascular events, i.e. the first occurrence of any of the following events: Death from any cause From cardiovascular causes From noncardiovascular causes Stroke or transitory ischemic attack (TIA) MI Hospitalization for repeat revascularization procedure, target (vessel) revascularization by means of PCI or CABG.

SECONDARY OUTCOMES:
Procedural success | 1 year
  The treatment will be considered successful when a complete hybrid revascularisation in the absence of complications during the index hospitalization has been achieved.
Pain assessment | 1 year
  assessment of visual analogue scale E.C. Huskisson

CONTACTS AND LOCATIONS:
Locations (1):
- A.V. Vishnevsky National Medical Research Center of Surgery., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No